CLINICAL TRIAL: NCT02813473
Title: SYNTAX III REVOLUTION Trial: A Randomized Study to Evaluate the Feasibility of Heart-Team Clinical Decision Making Regarding the Optimal (Surgical or Percutaneous Based) Revascularization Strategy in Patients With Complex Coronary Artery Disease, Based on Non-invasive Coronary CT Angiography (CTA) Imaging Utilising High-definition GE RevolutionTM Multi-slice CT and HeartFlow FFRCT Compared to the Current Standard of Care With Conventional Invasive Coronary Angiography (CA)
Brief Title: SYNTAX III REVOLUTION Trial: A Randomized Study Investigating the Use of CT Scan and Angiography of the Heart to Help the Doctors Decide Which Method is the Best to Improve Blood Supply to the Heart in Patients With Complex Coronary Artery Disease
Acronym: SYNTAX III
Status: Completed | Type: Observational
Sponsor: ECRI bv (Industry)
Collaborators: GE Healthcare (Industry); HeartFlow, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECRI-004
Record Dates: First submitted 2016-06-15; First posted 2016-06-27 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Diseases; Multivessel Coronary Artery Disease; Heart Diseases; Cardiovascular Diseases
Keywords: SYNTAX Score II; Multi Slice Computed Tomography; MSCT; Heart Team; Fractional Flow Reserve Computed Tomography; FFR; FFR MSCT; PCI; CABG; Percutaneous Coronary Intervention; Coronary Artery Bypass Graft
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Coronary Angiography — Coronary angiography is an X-ray test to diagnose diseases of the arteries that supply blood to the heart. Coronary angiography can detect weakened blood vessel walls and narrowed or blocked vessels. X-rays are taken after a special dye has been injected into the bloodstream, making the vessels and blood flow through the vessels visible on X-rays.
  Other Names: Angiogram; Coronary angiogram
Radiation: Computed Tomography (CT) scan — A CT scan is an X-ray imaging technique that uses a computer to produce cross-sectional images. It can be used to examine the heart and blood vessels for problems
  Other Names: Cardiac computed tomography; Multi-Slice CT scan (MSCT)

SUMMARY:
The SYNTAX III Revolution trial is a randomized diagnostic research study that investigates the use of CT scan and angiogram of the heart to help doctors decide which method is the best to improve blood supply to the heart in patients with complex coronary artery disease. Each patient will undergo an angiogram and CT scan per standard of care. The randomization strategy in this study is not between patients but between two teams of doctors, the so-called "Heart Teams", will be randomized: in the first round, team 1 assesses the angiogram, and team 2 assesses the CT scan. Then they make a decision about which treatment would be the best to treat complex coronary artery disease. In the second round, both teams see the imaging method that they did not see in the first round, and make the decision again. The final decision on the clinical treatment strategy is at the sole discretion of the Heart Team and there are no criteria described in SYNTAXIII Revolution protocol leading influencing this final decision.

Hypothesis: Determination of the best treatment strategy for coronary artery disease based on a CT scan will result in similar decisions as based on invasive coronary angiography.

DETAILED DESCRIPTION:
The SYNTAX III REVOLUTION Trial is a multicenter, all-comers trial (either isolated unprotected left-main or 3-vessel disease with or without left-main disease and candidate for either CABG or PCI treatment). In SYNTAXIII REVOLUTION a diagnostic coronary angiography and a diagnostic coronary Multislice CT are performed to allow the Heart Team to assess the optimal revascularization strategy. In a normal hospital setting the angiography is considered standard of care. The multislice CT can already also be part of the diagnosis and is at the discretion of the physician. After the images of both modalities are available, the patient will no longer participate in the trial. Next step is randomization of Heart Team A and Heart B to the sequence of availability of images, i.e. randomizing whether Heart Team A will review the angiography first or the multislice CT and, automatically, Heart B the other modality. The Heart Teams need to make a decision between surgical or percutaneous treatment according to either the conventional angiography or the multislice CT angiography assessment. In addition, the incremental value of FFRCT in the decision making of the Heart Team arm allocated primarily to the assessment of the MSCT (CT first algorithm) will be a secondary endpoint. No intervention to the patient's treatment takes place

i

ELIGIBILITY:
Inclusion Criteria:

1. Patients with at least 1 stenosis (angiographic, visually determined de novo lesions with ≥50% DS) in all 3 major epicardial territories (LAD and/or side branch, CX and/or side branch, RCA and/or side branch) supplying viable myocardium with or without left main involvement;
2. Patients with hypoplastic RCA with absence of descending posterior and presence of a lesion in the LAD and CX territories may be included in the trial as a 3VD equivalent;
3. Vessel size should be at least 1.5 mm in diameter as visually assessed in diagnostic angiogram;
4. Patients with chronic stable angina or stabilized acute coronary syndrome (inclusion criteria of the SYNTAX I study):

   * stable (Canadian Cardiovascular Society Class 1, 2, 3 or 4) angina pectoris;
   * or unstable (Braunwald class IB, IC, IIB, IIC, IIIB, IIIC) angina pectoris and ischemia with normal cardiac enzyme values prior to enrollment;
   * or patients with atypical chest pain or those who are asymptomatic provided they have myocardial ischemia (e.g. treadmill exercise test, radionuclide scintigraphy, stress echocardiography);
5. All anatomical SYNTAX Scores are eligible;
6. Patient amenable to a MSCT coronary angiography (e.g. no claustrophobia, high heartrate not amenable to beta-blockers, poor renal function, etc., up to discretion of investigator);
7. Patient has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Ethical Committee of the respective clinical site;

Exclusion Criteria:

1. Under the age of 18 years;
2. Unable to give Informed Consent;
3. Known pregnancy at time of enrolment. Female of childbearing potential (and last menstruation within the last 12 months), who are not taking adequate contraceptives. Female who is breastfeeding at time of enrolment;
4. Prior PCI or CABG; history of coronary stent implantation;
5. Evidence of evolving or ongoing acute myocardial infarction (AMI) in ECG and/or elevated cardiac biomarkers (according to local standard hospital practice) have not returned within normal limits at the time of enrollment;
6. Concomitant cardiac valve disease requiring surgical therapy (reconstruction or replacement);
7. Single or two-vessel disease (at time of Heart Team consensus);
8. Atrial fibrillation or significant arrhythmias;
9. Known allergy to iodinated contrast;
10. A Body Mass Index (BMI) of 35 or greater;
11. Participation in another trial with an investigational drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with complex coronary artery disease, defined as: left main (isolated, or associated with 1, 2 or 3 vessel disease) or de novo 3-vessel coronary artery disease (DS ≥50%), who are able to undergo cardiac CT with a GE high-definition RevolutionTM multi-slice CT scanner.
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W Serruys, Prof., Principal Investigator — Imperial College, London (UK)
Locations (6):
- BE006, Brussels, Belgium
- France (2):
  - FR013, Nancy
  - FR012, Paris
- DE011, Jena, Germany
- IT008, Milan, Italy
- CH003, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The research data will be entered on separate forms and stored under a code number, according to prevailing legal requirements. No names or other personal data will be stored. Only the study doctor will hold the information to link the code to the patients. The encoded data will be processed, analysed and reported by the research employees of this study, who have an obligation of secrecy.
  Representatives of the sponsor or members of the Ethics Committee (EC) and regulatory authorities within Europe can have access to the medical files in order to inspect the correctness of the research data. Data may be provided to representatives and affiliates of the industries supporting the study: General Electric and HeartFlow Inc. It is possible that the results of this study are presented or published in medical journals; this will always be without mention of the identity of the patients.

REFERENCES:
- [Derived] Andreini D, Modolo R, Katagiri Y, Mushtaq S, Sonck J, Collet C, De Martini S, Roberto M, Tanaka K, Miyazaki Y, Czapla J, Schoors D, Plass A, Maisano F, Kaufmann P, Orry X, Metzdorf PA, Folliguet T, Farber G, Diamantis I, Schonweiss M, Bonalumi G, Guglielmo M, Ferrari C, Olivares P, Cavallotti L, Leal I, Lindeboom W, Onuma Y, Serruys PW, Bartorelli AL; SYNTAX III REVOLUTION Investigators. Impact of Fractional Flow Reserve Derived From Coronary Computed Tomography Angiography on Heart Team Treatment Decision-Making in Patients With Multivessel Coronary Artery Disease: Insights From the SYNTAX III REVOLUTION Trial. Circ Cardiovasc Interv. 2019 Dec;12(12):e007607. doi: 10.1161/CIRCINTERVENTIONS.118.007607. Epub 2019 Dec 13. PMID 31833413
- [Derived] Collet C, Onuma Y, Andreini D, Sonck J, Pompilio G, Mushtaq S, La Meir M, Miyazaki Y, de Mey J, Gaemperli O, Ouda A, Maureira JP, Mandry D, Camenzind E, Macron L, Doenst T, Teichgraber U, Sigusch H, Asano T, Katagiri Y, Morel MA, Lindeboom W, Pontone G, Luscher TF, Bartorelli AL, Serruys PW. Coronary computed tomography angiography for heart team decision-making in multivessel coronary artery disease. Eur Heart J. 2018 Nov 1;39(41):3689-3698. doi: 10.1093/eurheartj/ehy581. PMID 30312411

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 223 patients with presence of 3 vessel dissease or left-main disease were enrolled in 6 centers in Europe to assess the coronary artery disease of the 223 patients randomized with either coronary CTA or conventional angiography blinded to the other modality.
Groups:
- Patients With Left Main or 3 Vessel Artery Disease: 223 patients with left main or 3 vessels artery desease were enrolled in the study. For each given patient the Heart Team is randomly assigned to an "Angio-First" or a "CT-First" decision algorithm. Each patient was assessed by both teams. The concordance or discordance of decision makings based on either conventional angiography (Angio first algorithm) or MSCT angiography (CT first algorithm) constitute the primary endpoint.
Period: Overall Study
Arm/Group | Patients With Left Main or 3 Vessel Artery Disease
Started | 223
Completed | 223
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With Left Main or 3 Vessel Artery Disease: Patients with left main or three-vessel coronary artery disease, diagnosed with either coronary CTA or conventional angiography and candidates for either CABG or PCI.
Arm/Group | Patients With Left Main or 3 Vessel Artery Disease
Number analyzed (Participants) | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 188
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Inter-rater Agreement on Revascularization Strategy of Two Heart Teams Using an "Angio-first" Algorithm or a "CT First" Algorithm.
Description: Inter-rater agreement, as assessed by Cohen's Kappa Kappa, on revascularization strategy of two Heart Teams using an "Angio-first" algorithm (based on invasive SYNTAX Score II) or a "CT-first" algorithm (based on non-invasive SYNTAX Score II, without FFRCT) and 95% confidence intervals (CI).
Time Frame: Heart Team meetings took place in average 1 to 2 weeks afer patient enrollment
Measure: Number (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Patients With Left Main or 3 Vessel Artery Disease
Number analyzed (Participants) | 223
proportion of agreement | 0.82 [0.73 to 0.91]

2. Secondary Outcome: Level of Agreement in the Decision Making Strategy Based on CT Only Without Functional Assessment and the Decision Making Strategy Based on CT With Functional Assessment ("CT First" Algorithm Group) at Screening.
Description: Analysis has not been done.
Time Frame: Nov 2017
Reporting Status: Not Posted

3. Secondary Outcome: Level of Agreement in the Decision Making Strategy Based on CT Only (With Functional Assessment) and the Decision Making Strategy Based on CT With Functional Assessment and Conventional Angiography ("CT First" Algorithm Group) at Screening
Description: Analysis has not been done.
Time Frame: Nov 2017
Reporting Status: Not Posted

4. Secondary Outcome: Level of Agreement in the Decision Making Strategy Based on Conventional Angiography Only and the Decision Making Strategy Based on CT With Functional Assessment and Conventional Angiography ("Angio First" Algorithm Group) at Screening
Description: Analysis has not been done.
Time Frame: Nov 2017
Reporting Status: Not Posted

5. Secondary Outcome: Inter-rater Agreement on Revascularization Strategy (Based on Conventional Angiography and CT With Functional Assessment) of Two Heart Teams Using an "Angio-first" Algorithm or a "CT-first" Algorithm at Screening
Description: Analysis has not been done.
Time Frame: Nov 2017
Reporting Status: Not Posted

6. Secondary Outcome: Anatomical SYNTAX Score Calculation Based on Non-invasive GE Revolution CT (Visual by Heart Team Involving an Experienced Coronary CT Reader) and the Resulting SYNTAX Score II at Screening
Description: Analysis has not been done.
Time Frame: Nov 2017
Reporting Status: Not Posted

7. Secondary Outcome: Anatomical SYNTAX Score Calculation Based on Non-invasive GE Revolution CT (Visual by Core Lab) and the Resulting SYNTAX Score II at Screening
Description: Analysis has not been done.
Time Frame: Nov 2017
Reporting Status: Not Posted

8. Secondary Outcome: Anatomical SYNTAX Score Calculation Based Invasive Angiography (Visual by Heart Team) and the Resulting SYNTAX Score II at Screening
Description: Analysis has not been done.
Time Frame: Nov 2017
Reporting Status: Not Posted

9. Secondary Outcome: Anatomical SYNTAX Score Calculation Based on Invasive Angiography (Visual by Core Lab) and the Resulting SYNTAX Score II at Screening
Description: Analysis has not been done.
Time Frame: Nov 2017
Reporting Status: Not Posted

10. Secondary Outcome: CT Based Functional Anatomy (FFRCT as Assessed by Heartflow) at Screening
Description: Analysis has not been done.
Time Frame: Nov 2017
Reporting Status: Not Posted

11. Secondary Outcome: Concordance in SYNTAX Score(s) Between and Within Strategies at Screening
Description: Analysis has not been done.
Time Frame: Nov 2017
Reporting Status: Not Posted

12. Secondary Outcome: Agreement in Coronary Stenosis Segments to be Revascularized Between and Within Strategies at Screening
Description: Analysis has not been done.
Time Frame: Nov 2017
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during patient participation in the study which started when informed consent was signed and ended when MSCT was done (if not available at the time of enrollment). That was between 1 and 5 days (max) from enrollement date.
Description: Patient participation started when informed consent was signed untill MSCT was done (if not available at the time of enrollment) between 1 and 5 days (max). Adverse events were collected in the study from first patient in until last patient MSCT that means 1 year and 8 months.
Arm/Group | Patients With Left Main or 3 Vessel Artery Disease
All-Cause Mortality (participants affected / at risk) | 0/223
Serious Adverse Events (participants affected / at risk) | 0/223
Other Adverse Events (participants affected / at risk) | 0/223

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT02813473/Prot_SAP_000.pdf